CLINICAL TRIAL: NCT01338675
Title: Targeted Busulfan, Fludarabine Conditioning Regimen for Hematopoietic Stem Cell Transplantation in Chronic Granulomatous Disease(CGD)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNUCH-SCT -1002
Record Dates: First submitted 2011-03-04; First posted 2011-04-19 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-11

CONDITIONS: Chronic Granulomatous Disease
Keywords: Chronic granulomatous disease; Hematopoietic Stem Cell Transplantation
MeSH Terms: conditions — Granulomatous Disease, Chronic | interventions — Busulfan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Busulfan (Experimental): First dose: busulfan (120 mg/m2 ivs once daily) (if age<1 yr: 80 mg/ m2) Second to forth dose: according to the daily pharmacokinetic study
  Interventions: Drug: Busulfan

INTERVENTIONS:
Drug: Busulfan — First dose: busulfan (120 mg/m2 ivs once daily) (if age<1 yr: 80 mg/ m2) Second to forth dose: according to the daily pharmacokinetic study

SUMMARY:
In this study the investigators plan to use optimal busulfan dose through pharmacokinetic study in stem cell transplantation of CGD patients.

DETAILED DESCRIPTION:
Chronic granulomatous disease is one of the rare congenital immunodeficiency which can be cured by hematopoietic stem cell transplantation. Previous myeloablative conditioning regimen has problems related to the severe toxicities, and non-myeloablative conditioning regimen has the risk of graft failure. Recently, reduced-intensity myeloablative conditioning regimen with busulfan and fludarabine was used usually in leukemia patients.

Busulfan is a highly toxic drug with narrow therapeutic window. In this study we plan to use optimal busulfan dose through pharmacokinetic study in stem cell transplantation of CGD patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are diagnosed as CGD.
* Patients who need hematopoietic stem cell transplantation with busulfan based conditioning regimen.
* Age: No limit.
* Performance status: ECOG 0-2.
* Patients must be free of significant functional deficits in major organs, but the following eligibility criteria may be modified in individual cases.
* Heart: a shortening fraction > 30% and ejection fraction > 45%.
* Liver: total bilirubin < 2 × upper limit of normal; ALT < 3 × upper limit of normal.
* Kidney: creatinine <2 × normal or a creatinine clearance (GFR) > 60 ml/min/1.73m2.
* Patients must lack any active viral infections or active fungal infection.
* Appropriate donor is available.
* Patients (or one of parents if patients age < 20) should sign informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2011-01; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Engraftment rate | 1 month after transplantation
  To evaluate engraftment rate after hematopoietic stem cell transplantation.

SECONDARY OUTCOMES:
Transplantation-related mortality and toxicities | 1, 3, 6 and 12 months after transplantation
  To evaluate 1-year event free survival after hematopoietic stem cell transplantation, toxicities associated with hematopoietic stem cell transplantation, acute and chronic GVHD, treatment related mortality and relapse rate.

CONTACTS AND LOCATIONS:
Overall Officials: Hyoung Jin Kang, M.D., Ph.D, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Daehangno, Jongno-gu, South Korea